CLINICAL TRIAL: NCT02543801
Title: A Prospective, Randomized Clinical Trial of Two Periarticular Multimodal Drug Injections in Total Hip and Knee Arthroplasty
Brief Title: A Clinical Trial of Two Periarticular Multimodal Drug Injections in Total Hip and Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kootenai Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB2022
Record Dates: First submitted 2015-08-21; First posted 2015-09-07 (Estimated); Results first posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Total Hip and Knee Arthroplasty
MeSH Terms: interventions — Ropivacaine; Bupivacaine; Clonidine; Ketorolac; Ketorolac Tromethamine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Hip Cohort Liposomal Bupivacaine (Active Comparator): Liposomal bupivacaine Bupivacaine Clonidine Epinephrine Ketorolac
  Interventions: Drug: Liposomal Bupivacaine; Drug: Bupivacaine; Drug: Clonidine; Drug: Ketorolac; Drug: Epinephrine
- Hip Cohort Ropivacaine (Active Comparator): Ropivacaine Clonidine Epinephrine Ketorolac
  Interventions: Drug: Ropivacaine; Drug: Clonidine; Drug: Ketorolac; Drug: Epinephrine
- Knee Cohort Liposomal Bupivacaine (Active Comparator): Liposomal bupivacaine Bupivacaine Clonidine Epinephrine Ketorolac
  Interventions: Drug: Liposomal Bupivacaine; Drug: Bupivacaine; Drug: Clonidine; Drug: Ketorolac; Drug: Epinephrine
- Knee Cohort Ropivacaine (Active Comparator): Ropivacaine Clonidine Epinephrine Ketorolac
  Interventions: Drug: Ropivacaine; Drug: Clonidine; Drug: Ketorolac; Drug: Epinephrine

INTERVENTIONS:
Drug: Liposomal Bupivacaine — Periarticular injection
  Other Names: Exparel
  Arms: Hip Cohort Liposomal Bupivacaine; Knee Cohort Liposomal Bupivacaine
Drug: Ropivacaine — Periarticular injection
  Other Names: Naropin
  Arms: Hip Cohort Ropivacaine; Knee Cohort Ropivacaine
Drug: Bupivacaine — Included as an element of the Liposomal bupivacaine intervention periarticular injection
  Other Names: Marcaine
  Arms: Hip Cohort Liposomal Bupivacaine; Knee Cohort Liposomal Bupivacaine
Drug: Clonidine — Included as an element of both interventions as a standard of care periarticular injection
  Other Names: Duraclon
Drug: Ketorolac — Included as an element of both interventions as a standard of care periarticular injection
  Other Names: Toradol
Drug: Epinephrine — Included as an element of both interventions as a standard of care periarticular injection
  Other Names: Adrenaline

SUMMARY:
This study evaluates two routinely used drug combinations for periarticular injection following total hip and knee arthroplasty for pain control. One group will receive liposomal bupivacaine, bupivacaine, clonidine, epinephrine and ketorolac. The other group will receive ropivacaine, clonidine, epinephrine and ketorolac.

DETAILED DESCRIPTION:
A key component of the multimodal approach to pain management is the intra-operative surgical site injection of a local anesthetic or drug cocktail. There are many formulations used for this purpose. A formulation documented in the literature was implemented by this institution which has dropped the average length of stay dramatically. Concern over the limited half-life of the administered anesthetic and the continued need for opioid administration has led to a search for better drug formulations and administration vehicles. Recently, the FDA approval of an extended release bupivacaine called liposomal bupivacaine was thought to extend the effective half-life of the anesthetic agent and thereby prolong post-operative anesthesia. Use of liposomal bupivacaine in total joint surgery was almost universally adopted after its recent approval and has been an integral part of the "same day total joint" movement.

Studies have suggested improvement in pain control and shortened hospitalizations with the use of liposomal bupivacaine. Other studies have raised questions about the effectiveness of this agent. Recently a randomized double blind study was performed with total knees which demonstrated no improvement in pain management with the addition of liposomal bupivacaine to the multimodal pain management protocol. This study has not been performed in the hip arthroplasty population.

ELIGIBILITY:
Inclusion Criteria:

* Hip Arthritis (osteoarthritis, post traumatic, inflammatory, and avascular necrosis)

Exclusion Criteria:

* Current use of opioid drugs
* Revision surgery
* Surgical complication (femoral fracture with implant insertion)
* Inability to provide Informed Consent

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe Bowen, MD, Principal Investigator — Kootenai Health

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hip Cohort: Enrollment began January 2016 and ended October 2017. Patients were recruited sequentially from a single orthopedic surgeon's practice.
  Knee Cohort: Enrollment began January 2017 and ended August 2018. Patients were recruited sequentially from three orthopedic surgeon practices.
Pre-assignment Details: Patients would be excluded if surgery was cancelled or for some clinical reason did not receive the periarticular injection during surgery.
Period: Overall Study
Arm/Group | Hip Cohort Liposomal Bupivacaine | Hip Cohort Ropivacaine | Knee Cohort Liposomal Bupivacaine | Knee Cohort Ropivacaine
Started | 61 | 60 | 59 | 59
Completed | 60 | 58 | 59 | 59
Not Completed | 1 | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hip Cohort Liposomal Bupivacaine | Hip Cohort Ropivacaine | Knee Cohort Liposomal Bupivacaine | Knee Cohort Ropivacaine | Total
Number analyzed (Participants) | 60 | 58 | 59 | 59 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (10) | 64 (11) | 66 (10) | 67 (9) | 66 (10)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: At the end of the study enrollment period 2 patients cancelled their surgeries and these were not replaced.
  Participants
    Female | 41 | 38 | 39 | 29 | 147
    Male | 19 | 20 | 20 | 30 | 89
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60 | 58 | 59 | 59 | 236

OUTCOME MEASURES:

1. Primary Outcome: Pain Score
Description: Self-reported pain score 0-10 (0=no pain - 10=worst possible pain experienced) and higher scores indicate a worse outcome
  Pain scores, collected every 4 hours per hospital care standards, were averaged (post-operatively up to 48 hours) to obtain individual mean pain scores and a mean score for the group was then calculated.
Time Frame: Starting post operatively and then every four hours up to 48 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hip Cohort Liposomal Bupivacaine | Hip Cohort Ropivacaine | Knee Cohort Liposomal Bupivacaine | Knee Cohort Ropivacaine
Number analyzed (Participants) | 60 | 58 | 59 | 59
score on a scale | 3.78 (2.22) | 3.85 (2.01) | 3.3 (2.0) | 3.4 (2.3)

2. Secondary Outcome: Narcotic Consumption
Description: Total amount of narcotics administered as calculated in oral morphine equivalent dose immediate post operatively up to 48 hours.
Time Frame: Starting immediately post operatively up to 48 hours
Measure: Mean (Standard Deviation); unit: morphine equivalents
Arm/Group | Hip Cohort Liposomal Bupivacaine | Hip Cohort Ropivacaine | Knee Cohort Liposomal Bupivacaine | Knee Cohort Ropivacaine
Number analyzed (Participants) | 60 | 58 | 59 | 59
morphine equivalents | 48.8 (22.9) | 57.4 (21.8) | 52.2 (28.4) | 50.0 (22.0)

3. Secondary Outcome: Length of Stay
Description: Measured in hours
Time Frame: Start of surgery to hospital discharge up to 140 hours
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Hip Cohort Liposomal Bupivacaine | Hip Cohort Ropivacaine | Knee Cohort Liposomal Bupivacaine | Knee Cohort Ropivacaine
Number analyzed (Participants) | 60 | 58 | 59 | 59
Hours | 33.8 (48.24655) | 50.3 (48.41333) | 36.0 (29.88427) | 38.4 (18.83953)

ADVERSE EVENTS:
Time Frame: Period of Hospitalization, began at end of surgery and ended at hospital discharge
Description: Because both arms are standard of care, adverse events would only be collected that did not relate to known and expected complications of surgery and total joint replacement.
Arm/Group | Hip Cohort Liposomal Bupivacaine | Hip Cohort Ropivacaine | Knee Cohort Liposomal Bupivacaine | Knee Cohort Ropivacaine
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/58 | 0/59 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/58 | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 0/60 | 0/58 | 0/59 | 0/59

LIMITATIONS AND CAVEATS:
Anesthesia (general or spinal) followed patient preference and not dictated by protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT02543801/Prot_SAP_000.pdf